CLINICAL TRIAL: NCT02325973
Title: Assessing Microvascular Resistance Via IMR To Predict Cumulative Outcome in STEMI Patients Undergoing Primary PCI (AMICRO)
Brief Title: Assessing Microvascular Resistance Via IMR To Predict Cumulative Outcome in STEMI Patients Undergoing Primary PCI
Acronym: AMICRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CV-12-018-IT-PW
Record Dates: First submitted 2014-01-30; First posted 2014-12-25 (Estimated); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Multi Vessel Coronary Artery Disease; STEMI
Keywords: STEMI; IMR; FFR; microcirculatory
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMR evaluation (Other): Assessment of IMR index in coronaries through PressureWire Certus guidewire
  Interventions: Device: PressureWire Certus guidewire

INTERVENTIONS:
Device: PressureWire Certus guidewire — Assessment of IMR index in coronaries through PressureWire Certus guidewire

SUMMARY:
The purpose of this study is to assess whether the Index of Microcirculatory Resistance (IMR) can be considered a prognostic predictor for the occurrence of events at one year of follow up after primary Percutaneous Coronary Intervention (PCI) in ST-Elevation Myocardial Infarction (STEMI) patients.

Any correlation between IMR and the short and medium term outcomes, defined as cardiovascular death, re-Myocardial Infarct (MI), re-hospitalization for Heart Failure (HF), resuscitation or Implantable Cardioverter Defibrillator (ICD) appropriate shock, will be assessed in the study.

DETAILED DESCRIPTION:
Prospective, multicentre study designed to evaluate IMR ability to predict events occurrence, defined as Cardiovascular death, re-MI, re-hospitalization for HF, resuscitation or ICD appropriate shock, during a 1 year follow-up period.

All participants will have the culprit lesion treated following clinical practice and guidelines; Fractional Flow Reserve (FFR) and IMR will be measured after the primary PCI procedure to evaluate treatment success and myocardial viability. Non-culprit lesions will be functionally evaluated through FFR index and will be treated if FFR will show functional stenosis. FFR and IMR will be measured to evaluate treatment success and myocardial viability. Patients will be followed-up at 1m, 6m and 1y periods.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of legal age in hosting country able and willing to provide informed consent form
2. Hospital admission either within 12 h of symptom onset or between 12 and 24 h after onset with evidence of continuing ischemia
3. Electrocardiographic ST-segment elevation ≥1 mm in two or more contiguous ECG leads, or with a left bundle-branch block (LBBB)
4. Multivessel diseased patients with lesions in the proximal 2/3 part of the vessels
5. Culprit Lesion EyeBall (EB) identified during evaluation of basal angiography
6. Presence of at least one non-culprit lesion >50% EB detected in the basal angiography and eligible for PCI for which the operators decision is to perform a staged pre-discharge angioplasty procedure

Exclusion Criteria:

1. Patients who cannot give informed consent
2. A life expectancy of less than 1 year
3. Patients who are pregnant or nursing
4. Contra-indication to angiography
5. Allergy/intolerance to Adenosine
6. Contra-indication/Allergy/Intolerance to contrast media or to medical therapy foreseen for PCI
7. Documented allergy to Adenosine diphosphate (ADP) inhibitors (aspirin and clopidogrel)
8. New infarct on the same area of a previous infarct
9. Critical non treatable Lesion EB>70% downstream of the culprit lesion
10. Absence of non-culprit lesion/s
11. Patient with hemodynamic instability not controllable with medical therapy and/or need intra aortic balloon pump implantation (IABP)
12. Prior Coronary Artery Bypass Graft (CABG) or indication for CABG
13. Patients with Left Main (LM) coronary artery disease requiring revascularization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2013-06; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Fineschi, MD, Study Chair — Policlinico Le Scotte, Siena; Marco Valgimigli, MD, Study Chair
Locations (14):
- Italy (14):
  - Ospedale Giovanni Paolo II, Sciacca, Agrigento
  - Ospedale Generale Regionale "F. Miulli", Acquaviva delle Fonti, BA
  - Azienda Ospedaliera Universitaria Careggi, Florence, FI
  - Azienda Ospedaliera Villa Scassi, Genova, GE
  - Fondazione Toscana G.Monasterio - Ospedale del Cuore, Massa, MS
  - Azienda Ospedaliera di Padova, Padua, PD
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro, PU
  - Fondazione IRCCS Policlinico S.Matteo, Pavia, PV
  - Arcispedale Santa Maria Nuova, Reggio Emilia, RE
  - Ospedale di Castelfranco Veneto, Castelfranco Veneto, Treviso
  - Presidio Ospedaliero di Conegliano, Conegliano, Treviso
  - Ospedale di Circolo Fondazione Macchi, Varese, VA
  - Ospedale Sant'Andrea, La Spezia
  - Policlinico Le Scotte, Siena

REFERENCES:
- [Derived] Fineschi M, Verna E, Barioli A, Mezzapelle G, Bartolini D, Turiano G, Guiducci V, Manari A, Lucarelli K, Uguccioni L, Repetto A, Tarantini G. One-year results from the Assessing MICRO-vascular resistances via IMR to predict outcome in ST-elevation myocardial infarction patients with multivessel disease undergoing primary PCI (AMICRO) trial. Front Cardiovasc Med. 2022 Dec 2;9:1051174. doi: 10.3389/fcvm.2022.1051174. eCollection 2022. PMID 36531736

RESULTS

PARTICIPANT FLOW:
Groups:
- STEMI Patient: STEMI patient treated with primary PCI with IMR evaluation. Study designed with 1 unique group
Period: Overall Study
Arm/Group | STEMI Patient
Started | 242
Completed | 221
Not Completed | 21
Not completed — Death | 5
Not completed — Withdrawal by subject or investigator | 16

BASELINE CHARACTERISTICS:
Arm/Group | IMR Evaluation
Number analyzed (Participants) | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 207
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] | 169.6 (6.9)
Weight [Mean (Standard Deviation); unit: kg] | 77 (11.8)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Normal range = 120-129 mmHg
  mmHg | 133.5 (24.8)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Normal range = 80-84 mmHg
  mmHg | 78.6 (13.8)
Heart Rate [Mean (Standard Deviation); unit: bpm (Beats Per Minute)] — Normal range = 60-100 bpm
  bpm (Beats Per Minute) | 74.5 (15.8)
Syntax Score (SS) [Mean (Standard Deviation); unit: units on a scale] — Measure of complexity grade of coronary artery disease; higher SS values indicate a more complex disease, a greater therapeutic challenge and potentially worse acute and long-term outcomes.
  SS categorization: score <= 22 -> low; score = 23-32 -> intermediate; score >= 33 -> high. Scale range: min score = 0; max score = 60
  units on a scale | 16.3 (5.8)
Infarcted area [Count of Participants; unit: Participants]
  Left Anterior Descending (LAD) coronary artery | 104
  Right Coronary Artery (RCA) | 100
  Circumflex Artery (CX) | 38
Participants with Hypertension [Count of Participants; unit: Participants] | 116
Participants with Diabetes [Count of Participants; unit: Participants]
  Diet | 5
  Insulin | 7
  Oral treatment | 25
  None | 205
Parrticipants with Hyperlipidemia and/or Dyslipidemia [Count of Participants; unit: Participants] | 105
Participants with Renal dysfunction [Count of Participants; unit: Participants]
  Without dialysis | 3
  With dialysis | 0
  None | 239
Participants with significant alcohol intake [Count of Participants; unit: Participants] | 3
Smoker [Count of Participants; unit: Participants]
  Current | 100
  Ex smoker | 31
  None | 111
Participants with history of stroke [Count of Participants; unit: Participants] | 3
Participants with history of Transient Ischemic Attach (TIA) [Count of Participants; unit: Participants] | 5
Participants with history of Myocardial Infarction [Count of Participants; unit: Participants] | 7
Participants with history of Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants] | 13
Participants with Family history of heart disease [Count of Participants; unit: Participants] | 67
Participants with history of Heart failure [Count of Participants; unit: Participants] | 3
Killip class [Count of Participants; unit: Participants] — Higher class means patient more compromise. Class 1: Absence of rales over the lung fields and absence of a third heart sound (S3) Class 2: Rales over 50% or less of the lung fields or the presence of an S3 Class 3: Rales over more than 50% of the lung fields Class 4: Cardiogenic Shock
  Participants
    Class I | 230
    Class II | 12
    Class III | 0
    Class IV | 0

OUTCOME MEASURES:

1. Primary Outcome: Composite of: Cardiovascular Death*, Re-myocardial Infarct, Re-hospitalization for Heart Failure (HF) and Congestive Heart Failure (CHF), Resuscitation or ICD Appropriate Shock.
Description: Composite of: cardiovascular death*, re-myocardial infarct, re-hospitalization for heart failure (HF) and Congestive Heart Failure (CHF), resuscitation or ICD appropriate shocK, at 1 year.
  * = timing of mortality evaluation: once culprit lesion has been evaluated through IMR
  Composite endpoint was evaluated as time to first event, whichever individual component occurred first.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | STEMI Patient
Number analyzed (Participants) | 242
Participants | 8

2. Secondary Outcome: New Congestive Heart Failure (CHF) During Index Hospitalization
Description: Count of participants with a new CHF during index hospitalization. Hospital stay expected average = 5-10 days
Time Frame: At the end of hospital stay
Population: Participants that had a new congestive heart failure (CHF) during index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | STEMI Patient
Number analyzed (Participants) | 242
Participants | 8

3. Secondary Outcome: Left Ventricular (LV) Remodeling
Description: Left Ventricular (LV) remodeling at 1 year; improvement of Ejection Fraction %(EF) assessed by TTE.
  A TTE evaluation has been done both at discharge and at 1-year fup.
Time Frame: 1 year
Population: Echo data site reported, a complete echo has not been always done during discharge and fup visits.
Measure: Mean (Standard Deviation); unit: % of ejection fraction
Groups:
- STEMI Pat. at Discharge: ECHO DISCHARGE EVALUATION
- STEMI Pat. at 1 Y Fup: 1 YEAR FOLLOW EVALUATION
Arm/Group | STEMI Pat. at Discharge | STEMI Pat. at 1 Y Fup
Number analyzed (Participants) | 202 | 202
% of ejection fraction | 53.3 (8.6) | 56.2 (7.9)

4. Secondary Outcome: Left Ventricular (LV) Remodeling
Description: Left Ventricular (LV) remodeling at 1 year; improvement of Left Ventricular End Systole Volume (LVESV) and Left Ventricular End Diastole Volume (LVEDV) assessed by TTE.
  A TTE evaluation has been done both at discharge and at 1-year fup.
Time Frame: 1 year
Population: Echo data site reported, a complete echo has not been always done during discharge and fup visits.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | STEMI Pat. at Discharge | STEMI Pat. at 1 Y Fup
Number analyzed (Participants) | 191 | 191
ml
  LVESV (ml): number analyzed (Participants) | 190 | 190
  LVESV (ml) | 50.6 (21.8) | 47.4 (20.3)
  LVEDV (ml) | 101.7 (28.5) | 102.3 (32.4)

5. Secondary Outcome: Left Ventricular (LV) Remodeling
Description: Left Ventricular (LV) remodeling at 1 year; improvement of Left Ventricular End Diastole Diameter (LVEDD) and Left Ventricular End Systole Diameter (LVESD) assessed by TTE.
  A TTE evaluation has been done both at discharge and at 1-year fup.
Time Frame: 1 year
Population: Echo data site reported, a complete echo has not been always done during discharge and fup visits.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | STEMI Pat. at Discharge | STEMI Pat. at 1 Y Fup
Number analyzed (Participants) | 182 | 182
mm
  LVESD (mm): number analyzed (Participants) | 168 | 168
  LVESD (mm) | 35.5 (8.5) | 33.9 (6.6)
  LVEDD (mm) | 51.4 (29.7) | 50.2 (7.5)

6. Secondary Outcome: Left Ventricular (LV) Remodeling
Description: Left Ventricular (LV) remodeling at 1 year; improvement of 16 segments Wall Motion Score Index (WMSI) assessed by TTE.
  A TTE evaluation has been done both at discharge and at 1-year fup. 16WMSI = 1 is considered normokinetic; 16WMSI = 1,5 is considered mild hypokinesia; 16WMSI = 2 is considered hypokinesia; 16WMSI = 2,5 is considered severe hypokinesia; 16WMSI = 3 is considered akinetic.
  Scale range: from 1 to 3
Time Frame: 1 year
Population: Echo data site reported, a complete echo has not been always done during discharge and fup visits.
Measure: Mean (Standard Deviation); unit: index
Arm/Group | STEMI Pat. at Discharge | STEMI Pat. at 1 Y Fup
Number analyzed (Participants) | 195 | 195
index | 1.8 (2.9) | 1.9 (3.9)

7. Secondary Outcome: Left Ventricular (LV) Remodeling - Mitral Insufficiency
Description: Left Ventricular (LV) remodeling at 1 year; improvement of mitral insufficiency (MI) values assessed by TTE.
  A TTE evalutation has been done both at discharge and at 1-year fup. Each row reports the number of participants that have that specific grade of mitral insufficiency.
  Grade = 0 indicates no MI; grade = 1 indicates mild MI; grade = 2 indicates moderate MI; grade = 3 indicates severe MI
Time Frame: 1 year
Population: Echo data site reported, a complete echo has not been always done during discharge and fup visits
Measure: Count of Participants; unit: Participants
Arm/Group | STEMI Pat. at Discharge | STEMI Pat. at 1 Y Fup
Number analyzed (Participants) | 199 | 199
Participants
  Grade 0 | 35 | 33
  Grade 1 | 130 | 139
  Grade 2 | 29 | 26
  Grade 3 | 5 | 1

8. Secondary Outcome: Need for New Revascularization
Description: Incidence of new revascularizations at 1 year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | STEMI Patient
Number analyzed (Participants) | 242
Participants | 12

9. Secondary Outcome: Stent Thrombosis
Description: Incidence of stent thrombosis at 1 year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | STEMI Patient
Number analyzed (Participants) | 242
Participants | 1

10. Secondary Outcome: Evaluation of a Better Cut-off of IMR Index Based on Primary Endpoints Events
Description: Evaluation of a better cut-off of IMR index based on primary endpoints events. Table below reports the values of ROC curve.
Time Frame: 1 year
Measure: Number; unit: probability
Groups:
- True Positive Rate: True positive rate, data related to post primary IMR measurement
- False Positive Rate: False positive rate, data related to post primary IMR measurement
- Area Under the Curve: Area under the curve, data related to post primary IMR measurement
Arm/Group | True Positive Rate | False Positive Rate | Area Under the Curve
Number analyzed (Participants) | 242 | 242 | 242
probability
  IMR cut-off value = 95 | 0.125 | 0.114 | 0.505
  IMR cut-off value = 65 | 0.375 | 0.211 | 0.582
  IMR cut-off value = 55 | 0.5 | 0.281 | 0.610
  IMR cut-off value = 48 | 0.625 | 0.325 | 0.650
  IMR cut-off value = 34.5 | 0.75 | 0.491 | 0.629
  IMR cut-off value = 32 | 0.875 | 0.531 | 0.672
  IMR cut-off value = 30 | 0.875 | 0.57 | 0.652
  IMR cut-off value = 20 | 0.875 | 0.768 | 0.554

11. Secondary Outcome: Evaluation of Possible Events Predictors
Description: Results of logistic regression model; differences were considered statistically significant when p<0,05.
Time Frame: 1 year
Measure: Number; unit: correlation coefficient
Arm/Group | STEMI Patient
Number analyzed (Participants) | 242
correlation coefficient
  Age | 0,3139
  Male | 0,8407
  Number of PCIs (PCIs done both during Primary and Staged procedures) | 0,0415
  Hypertension | 0,3039
  Lipids | 0,1948
  Smoking | 0,5603
  LVEF (at discharge) | 0,0320
  WMSI (at discharge) | 0,2320

ADVERSE EVENTS:
Time Frame: Adverse event data have been collected over 1 year period of time from primary procedure
Arm/Group | STEMI Patient
All-Cause Mortality (participants affected / at risk) | 5/242
Serious Adverse Events (participants affected / at risk) | 58/242
Other Adverse Events (participants affected / at risk) | 16/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STEMI Patient (N=242)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Angina or atypical chest pain (Cardiac disorders) | 3 (3)
Asystolia (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 3 (3)
Planned ICD implantation for primary disease (Cardiac disorders) | 1 (1)
COPD reacutization (Cardiac disorders) | 1 (1)
Effort angina (Cardiac disorders) | 2 (2)
Heart failure (Cardiac disorders) | 5 (5)
Iatrogenic sinus bradycardia (Cardiac disorders) | 1 (1)
Coronary revascularization (Cardiac disorders) | 5 (5)
Planned angiography (Cardiac disorders) | 1 (1)
Mitral regurgitation (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 2 (2)
Pulmonary stasis (Cardiac disorders) | 1 (1)
Parossistic dyspnoea (Cardiac disorders) | 1 (1)
Stable angina (Cardiac disorders) | 2 (2)
Bleeding from duodenal angiodysplasia (Gastrointestinal disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1)
Planned angiography for control (Investigations) | 1 (1)
Broken femur (Musculoskeletal and connective tissue disorders) | 1 (1)
Ischaemic (Nervous system disorders) | 1 (1)
TIA in left side with right hemiparesis (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Iatrogenic syncope (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary Sepsi (Renal and urinary disorders) | 2 (2)
Kidney insufficiency (Renal and urinary disorders) | 1 (1)
Fever, possible pleuritis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung neoplasia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intra-stent thrombosis (Vascular disorders) | 3 (3)
Coronary artery dissection (Vascular disorders) | 3 (3)
Femoral hematoma (Vascular disorders) | 1 (1)
Thrombosis of radial right forearm (Vascular disorders) | 1 (1)
Cardiogenic shock (Vascular disorders) | 1 (1)
Right femoral region leakage (Vascular disorders) | 1 (1)
Hypotensive syncope betablocker related (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STEMI Patient (N=242)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Chest pain (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Probably neuralgic pain (Nervous system disorders) | 1 (1)
Lypothymia (Nervous system disorders) | 1 (1)
Chest pain not coronary related (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cought (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asymptomatic culprit vessel occlusion founded during staged procedure (Vascular disorders) | 1 (1)
Acute thrombosis stent (Vascular disorders) | 1 (1)
Astenia, hypotension (Vascular disorders) | 1 (1)
Epistaxis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Since it is a multicenter study,no results presentation or publication shall be made prior to the communication,presentation or publication to congresses and/or scientific journals without Sponsor consent.Investigator has to provide copy of any proposed Publication&all related materials to Sponsor for consideration at least 30 days prior to the proposed submission date.Sponsor can ask Investigator to refrain from making the Publication for 60 days in order to verify the accuracy of information

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT02325973/Prot_SAP_000.pdf